CLINICAL TRIAL: NCT00641134
Title: Cardiac Rehabilitation in Advanced aGE: EXercise TRaining and Active Follow-up, a Randomised Controlled Trial. CR-AGE EXTRA Trial
Brief Title: Cardiac Rehabilitation in Advanced aGE: EXercise TRaining and Active Follow-up CR-AGE-EXTRA Trial
Acronym: CR-AGE-EXTRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Florence (Other)
Responsible Party: Francesco Fattirolli, MD, PhD, Azienda Ospedaliero-Universitaria Careggi - Florence, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 93/2007
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Cardiovascular Disease
Keywords: Cardiac Rehabilitation; Old age; Home physical training
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): A:Home-Based exercise program,-at discharge from in-Hospital CR program-, with one reinforcement session each month for the first 6 months.
  Interventions: Other: A: Home-Based exercise after Cardiac Rehabilitation
- B (No Intervention): Usual care, after CR, consisting of recommendation on usefulness of physical exercise and standard follow-up visits and functional assessment at 6 and 12 months.

INTERVENTIONS:
Other: A: Home-Based exercise after Cardiac Rehabilitation — Home-Based exercise program,after CR, with reinforcement sessions
  Other Names: Home-based exercise after CR
  Arms: A

SUMMARY:
The goal of this trial is to assess the medium- (6 months) and long-term (12 months) effects of a Home-Based exercise program after in-Hospital comprehensive Cardiac Rehabilitation (CR) - as compared with usual care - on exercise capacity, health-related quality of life and health care services utilization, in patients (pts) older than 75 years after recent acute coronary syndromes or cardiac surgery.

DETAILED DESCRIPTION:
Data on the short-term efficacy of comprehensive CR are still limited in older pts with cardiovascular disease, and no information is available on maintenance of results achieved with CR over the medium- and long-term periods. As long-term adherence with exercise programs after comprehensive CR is generally poor, with only 30% reporting regular exercise at 12-month follow-up, guidelines recommend the implementation of methods aimed at improving adherence with such programs. The applicability to older pts of Home-Based exercise programs aimed at enhancing the adherence with prescriptions and maintaining the physiological benefits attained during the in-Hospital training period, is a further issue still to be clarified. The goal of this study is to determine in pts older than 75 years the medium- (6 months) and long-term (12 months) effects of a Home-Based exercise program after in-Hospital comprehensive CR, as compared with usual care, on exercise capacity, health-related quality of life and health care services utilization.

Pts older than 75 years who are candidate to an in-Hospital comprehensive CR program after acute coronary syndromes (ACS), percutaneous coronary intervention (PCI) or cardiac surgery (coronary artery by-pass graft and/or valvular surgery), will be screened for eligibility in the trial, and will be enrolled provided they do not meet any of the exclusion criteria. At baseline, at completion of CR program, and at 6- and 12-month follow-up, the following data will be assessed in all enrolled pts:

* functional capacity, expressed as total work capacity (TWC, watt) and maximal aerobic capacity (peak VO2, ml/kg/min) during a symptom-limited cardiopulmonary exercise test
* endurance, expressed by the distance covered during a 6-minute walk test (6MWT)
* lower limb muscular strength, measured with an isokinetic dynamometer
* health-related quality of life (SF 36 questionnaire)
* utilization rates of health care services

At discharge from in-Hospital CR program, pts will be randomly allocated to:

1. Home-Based exercise program, consisting of a prescription of a specific set of exercises detailed and actively recorded in a log book, with one reinforcement session at the Rehabilitation Centre each month for the first 6 months.
2. Usual care, consisting of recommendation on usefulness of physical exercise and standard follow-up visits and functional assessment at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Women and men
* Aged >75 years
* Candidates to a 4-week
* In-Hospital comprehensive CR after ACS
* PCI
* Cardiac surgery

Exclusion Criteria:

* Any medical condition that would make physical exercise unsafe (unstable angina, sustained ventricular arrhythmias, AF with elevated ventricular response, symptomatic COPD, uncontrolled arterial hypertension, uncontrolled diabetes, hyperthyroidism) or that would limit physical capacity (severe anemia (Hb<10 gr/dl), moderate-to-severe chronic renal failure (creatinine >2.5 mg/dl), severe arthritis, peripheral artery disease (Fontaine >IIb), metastatic cancer)
* Symptomatic (NYHA II-IV) chronic heart failure
* Moderate-to-severe left ventricular systolic dysfunction (left ventricular ejection fraction <35%)
* BADL disability
* Denied informed consent

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
functional capacity at 6- and 12-months after CR in pts older than 75 years randomly allocated to Home-Based exercise program or usual care. | 6 and 12 months

SECONDARY OUTCOMES:
health-related quality of life and health care services utilization rates. | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Fattirolli, MD, PhD, Study Director — Azienda Ospedaliero-Universitaria Careggi - Florence, Italy
Locations (1):
- Azienda Ospedaliero-Universitaria Careggi - Florence, Florence, Italy

REFERENCES:
- [Derived] Pratesi A, Baldasseroni S, Burgisser C, Orso F, Barucci R, Silverii MV, Venturini S, Ungar A, Marchionni N, Fattirolli F. Long-term functional outcomes after cardiac rehabilitation in older patients. Data from the Cardiac Rehabilitation in Advanced aGE: EXercise TRaining and Active follow-up (CR-AGE EXTRA) randomised study. Eur J Prev Cardiol. 2019 Sep;26(14):1470-1478. doi: 10.1177/2047487319854141. Epub 2019 Jun 10. PMID 31180763